CLINICAL TRIAL: NCT01726296
Title: Adherence to NCCN Survivorship Care Guidelines in Non-Small Cell Lung Cancer and Colorectal Cancer Survivor Care
Brief Title: Adherence to Survivorship Care Guidelines in Health Care Providers for Non-Small Cell Lung Cancer and Colorectal Cancer Survivor Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 12-841; NCI-2012-01717 (Registry Identifier: NCI CTRP Registration Site)
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2016-11

CONDITIONS: Adenocarcinoma of the Lung; Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Squamous Cell Lung Cancer; Stage I Colon Cancer; Stage I Rectal Cancer; Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer; Stage IIA Colon Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIA Rectal Cancer; Stage IIB Colon Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIB Rectal Cancer; Stage IIC Colon Cancer; Stage IIC Rectal Cancer; Stage IIIA Colon Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Colonic Neoplasms; Rectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health services research (educational intervention) (Experimental): Health care providers complete an educational intervention based on NCCN guidelines in CRC and NSCLC survivorship care comprising a power point presentation reviewing evidence and prompts for addressing survivorship care components; and an electronic paper copy sample survivorship care plan that can be adapted and distributed at each participating site.
  Interventions: Other: educational intervention; Other: medical chart review

INTERVENTIONS:
Other: educational intervention — Complete an educational intervention based on NCCN guidelines and disease-specific issues related to survivorship care
  Other Names: intervention, educational
Other: medical chart review — Complete patient medical chart audit
  Other Names: chart review

SUMMARY:
This clinical trial studies adherence to survivorship care guidelines in health care providers for non-small cell lung cancer or colorectal cancer survivor care. The completion of an educational intervention by health care providers may increase compliance and adherence to National Comprehensive Cancer Network guidelines for survivorship care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate adherence of oncology health care providers to National Comprehensive Cancer Network (NCCN) guidelines for cancer survivorship care in colorectal cancer (CRC) and non-small cell lung cancer (NSCLC) cancers.

SECONDARY OBJECTIVES:

I. To develop and assess a targeted educational initiative to improve compliance with NCCN CRC and NSCLC survivorship guidelines for oncology health care providers in academic and community practice.

II. To evaluate the impact of this educational initiative on documented adherence and compliance with NCCN guidelines for NSCLC and CRC survivorship care by oncology health care providers.

OUTLINE:

Health care providers complete an educational intervention based on NCCN guidelines in CRC and NSCLC survivorship care comprising a power point presentation reviewing evidence and guidelines; a USB drive of the NCCN guidelines with paper copy of pages addressing survivorship care; an electronic and paper copy of a sample survivorship clinic template note with prompts for addressing survivorship care components; and an electronic paper copy sample survivorship care plan that can be adapted and distributed at each participating site.

ELIGIBILITY:
Inclusion Criteria:

* HEALTH CARE PROVIDER INCLUSION CRITERIA:
* Any health care provider (physician, advanced practice clinician) at a study site (Fox Chase Cancer Center [FCCC] and Fox Chase Cancer Center Partners [FCCCP]) who provides care for NSCLC and/or CRC survivors
* CHART AUDIT INCLUSION CRITERIA (BASELINE):
* Cancer Registry cases include stage I-III colon cancer (adenocarcinoma histology), stage I-III rectal cancer (adenocarcinoma histology), stage I-III non-small cell lung cancer (squamous or adenocarcinoma histology)
* Patients must have completed all therapy for curative intent at least six months prior to chart audit
* Undergoing routine oncology care and surveillance at the chosen site (defined as receiving follow-up care with FCCC or FCCCP site health care providers and have an active medical chart)
* No evidence of metastatic disease
* Patients must have been seen for a visit for cancer surveillance between 2009 and 2013
* Health care providers at the participating site must be willing and able to participate in the educational initiative
* CHART AUDIT INCLUSION CRITERIA (POST-INTERVENTION)
* Charts eligible for audit after completion of the educational initiative will be for those CRC and NSCLC survivors presenting for follow-up after the initiative has been completed by site health care providers

Exclusion Criteria:

* CHART AUDIT EXCLUSION CRITERIA:
* Cancer Registry cases for diseases other than colon or rectal adenocarcinoma and non-small cell lung cancer (squamous or adenocarcinoma histology)
* Patients currently receiving active therapy for any cancer, including CRC or NSCLC
* Patients who do not undergo routine oncologic care at the chosen Partners site or Fox Chase Cancer Center
* Stage IV cancer or evidence of metastatic disease at any time point
* Patients who have not undergone a visit for cancer surveillance since 2009
* Fox Chase Cancer Partners sites who do not agree to chart audit procedures or providers are unable or unwilling to participate in the educational initiative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Percentage of eligible CRC and NSCLC survivors with medical record documentation of compliance with NCCN guidelines | Up to 6 months
  A test of the binomial proportion will have 99% power with 1% type I error to make this distinction.

SECONDARY OUTCOMES:
Change in percentage of eligible survivors with documentation of compliance with NCCN survivorship guidelines after conducting the targeted educational initiative at participating sites | Baseline and up to 6 months
  This two-sample test of binomial proportions will have 99% power with 1% type I error.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Denlinger, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States